CLINICAL TRIAL: NCT06188039
Title: Predicting Fluid REsponsiveness Using Superior Vena Cava Collapsibility IndEx duriNg High-risk Non-Cardiac surgEry (PRESCIENCE)
Brief Title: Superior Vena Cava Collapsibility Index for Predicting Fluid Responsiveness During High-risk Non-cardiac Surgery
Acronym: PRESCIENCE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Uniwersytecki Szpital Kliniczny w Opolu (Other)
Responsible Party: Principal Investigator, Tomasz Królicki, MD PhD, Principal Investigator, Uniwersytecki Szpital Kliniczny w Opolu
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: W27/KB/2023_TK
Record Dates: First submitted 2023-12-13; First posted 2024-01-03 (Actual); Last update posted 2026-01-06 (Actual); Status verified 2024-01

CONDITIONS: Surgery; Fluid Responsiveness; Transesophageal Echocardiography
Keywords: Fluid responsiveness; non-cardiac surgery; Superior vena cava collapsibility index; echocardiography
MeSH Terms: interventions — Echocardiography, Transesophageal

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Patients undergoing open aortic surgery with sinus rhythm (Experimental): Arm to validate SVC-CI during open aortic surgery with special focus of predicting FR during aortic cross clamping (n=50).
  Interventions: Diagnostic Test: Superior vena cava collapsibility index
- Patients undergoing laparotomy and high PEEP (Experimental): Arm designed to validate SVC-CI during laparotomy, ventilated with high PEEP levels (8-10cmH2O). PEEP will be raised transiently during measurements (n=50).
  Interventions: Diagnostic Test: Superior vena cava collapsibility index; Other: PEEP elevation
- Patients undergoing laparotomy with standard ventilatory settings (Active Comparator): Arm designed as an active comparator with standard (protective) ventilatory settings (n=50). Tidal volumes (Vt) will be set for 8ml/kg.
  Interventions: Diagnostic Test: Superior vena cava collapsibility index

INTERVENTIONS:
Diagnostic Test: Superior vena cava collapsibility index — After induction of general anaesthesia following interventions will be performed.
  1. Insertion of a tranesophageal echocardiography probe
  2. Measurement of SVC-CI
  3. Measurement of LVOT-VTI prior to fluid bolus
  4. Fluid bolus (250ml of crystalloid)
  5. Measurement of LVOT-VTI after fluid bolus
  Several volume trials per patient will be allowed, until safety criteria are met. In such cases further testing will be stopped.
  Other Names: SVC-CI; fluid bolus; transesophageal echocardiography
Other: PEEP elevation — A transient elevation of positive end-expiratory pressure (PEEP) will be applied, in order to validate SVC-CI in the setting of elevated PEEP.
  A PEEP level of 8-10cmH2O will be applied for 1 minute prior to every measurement of SVC-CI. Then the previous PEEP level will be reinstated.
  Arms: Patients undergoing laparotomy and high PEEP

SUMMARY:
The goal of this prospective study is to validate the superior vena cava collapsibility index (SVC-CI) as a predictor of fluid responsiveness during laparotomy and open aortic surgery. The SVC-CI and patients' response to fluid will be assessed based on transesophageal echocardiography.

The study has three arms, in order to validate SVC-CI under the conditions of laparotomy, aortic cross clamping and high PEEP levels. One of the study arms will be an active comparator arm.

The data obtained from this study may help physicians guide intraoperative fluid therapy in a more efficient manner, in order to decrease perioperative mortality.

DETAILED DESCRIPTION:
Patients undergoing high-risk non-cardiac surgery, including acute laparotomies and open aortic surgery, are at high risk of postoperative complications and adverse cardiovascular events. Perioperative fluid therapy is a factor which is strongly associated with postoperative outcomes. To avoid both hypovolemia and excessive fluid administration a strategy of goal-directed fluid therapy (GDFT) has been coined. Traditionally in the setting of operating rooms GDFT relied on stroke-volume variation (SVV) measured by hemodynamic monitors, based on uncalibrated pulse contour cardiac output analysis (uAPCO). However in the described cohort of patients uAPCO methods show a significantly increased measurement error, which is mainly attributed to dynamic changes in peripheral vascular tone. Furthermore, frequent occurrence of arhytmias in those patients limits the use of SVV and all other dynamic indices of fluid responsiveness based on those methods. Superior vena cava collapsibility index (SVC-CI) is a parameter which is devoid of the above mentioned limitations. It relies on respiratory variation of superior vena cava during the respiratory cycle and is therefore reliable in patients with irregular heart rhytm and seems independent from changing afterload conditions.

The main purpose of this study is to validate SVC-CI in patients undergoing controlled mechanical ventilation during laparotomies and during open aortic surgery, with focus on elevated PEEP levels and aortic cross-clamping.

ELIGIBILITY:
Inclusion Criteria:

* Signed ICF (informed consent form)
* Age > 18 years old Eligibility criteria for each arm (additionally to mandatory criteria)
* Arm 1 - Patients undergoing open aortic surgery
* Arm 2 - Patients undergoing laparotomy
* Arm 3 - Patients undergoing laparotomy with sinus rhytm

Exclusion Criteria:

1. Patients who are deemed to be at risk of harm due to excessive fluid administration:

   * End-stage renal disease (eGFR <15ml/kg/min)
   * Decompensated heart failure
   * Respiratory failure prior to surgery
   * Other cases where the risk of harm from fluid overload is assessed to be significant by the investigator
2. Medical contraindication to the use of transesophageal echocardiography:

   * Active ulcerative gastritis or bleeding from upper gastrointestinal tract
   * Past history of esophageal or gastric surgery
   * Esophageal varices or other esophageal disease (stricture, Barret's disease, perforation in the past, achalasia)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2024-01-03 (Actual); Primary Completion 2025-11-17 (Actual); Study Completion 2025-11-18 (Actual)

PRIMARY OUTCOMES:
Fluid responsiveness | Directly after infusing fluid bolus.
  Fluid responsiveness was defined as an increase of 10% or more of cardiac output (CO) following an administered 250ml fluid bolus. Changes in CO will be estimated using changes in left ventricle outflow tract velocity time integral (LVOT-VTI) assessed by transesophageal echocardiography to avoid errors associated with measuring LVOT area, which is necessary to calculate CO.

CONTACTS AND LOCATIONS:
Overall Officials: Tomasz Królicki, MD, PhD, Study Chair — Uniwersytecki Szpital Kliniczny w Opolu
Locations (1):
- Opole University Hospital, Opole, Poland

IPD SHARING:
Plan to Share IPD: No
The data will be shared in open access, however no plan has been designed.